CLINICAL TRIAL: NCT00491686
Title: A Phase IIa, Multi-Center, Randomized, Double-blind, Placebo-controlled, Parallel-Group Study to Assess the Antidepressant Effect and Onset of Effect of AZD6765 in Treatment-Resistant Major Depressive Disorder Patients
Brief Title: AZD6765 for Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD - Emerging Psychiatry Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6702C00001
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Depression
Keywords: Long-term depression
MeSH Terms: conditions — Depression | interventions — AZD6765

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: AZD6765 — intravenous infusion

SUMMARY:
The purpose of this study is to determine whether treatment with AZD6765 will have an antidepressant effect with patients who have treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Depression
* Inadequate response to an adequate course of antidepressants

Exclusion Criteria:

* Psychiatric disorder other than depression
* Pregnancy or lactation
* Current diagnosis of cancer

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine whether an antidepressant effect can be achieved in patients with Treatment Resistant Depression determined by a change from baseline in the MADRS total score. | Change from Baseline

SECONDARY OUTCOMES:
The secondary objective is to assess the safety and tolerability of AZD6765 as assessed by vital signs, physical examination, clinical laboratory evaluations, ECG's and incidence of adverse events. | each visit; change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mark Smith, MD, PhD, Study Director — AstraZeneca
Locations (5):
- United States (5):
  - Research Site, Glendale, California
  - Research Site, Hartford, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Wichita, Kansas
  - Research Site, Rockville, Maryland

REFERENCES:
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Sanacora G, Smith MA, Pathak S, Su HL, Boeijinga PH, McCarthy DJ, Quirk MC. Lanicemine: a low-trapping NMDA channel blocker produces sustained antidepressant efficacy with minimal psychotomimetic adverse effects. Mol Psychiatry. 2014 Sep;19(9):978-85. doi: 10.1038/mp.2013.130. Epub 2013 Oct 15. PMID 24126931